CLINICAL TRIAL: NCT04484662
Title: Effects of Potted Mint Plants on Indoor Air Quality and the Concentration of Bacterium and Fungus, and Evaluation of Cardiovascular Health
Brief Title: Potted Mint Plants
Acronym: PMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 202005078RIND
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-07

CONDITIONS: Cardiovascular Diseases
Keywords: Potted mint plants; Indoor air quality; Fungus; Bacteria; Cardiovascular health
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This study will recruit 60 subjects, in sum of 30 families.
Masking Description: This study will recruit 60 subjects, in sum of 30 families.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Potted Mint Plants Intervention (Other): We will measure 2 indoor environments (living room and bedroom) for placing potted plants. We will analyze the effect of potted mint plants on indoor air quality, fungal and bacterial concentration, and explore the correlation between the intervention of potted mint plants and cardiovascular health.
  Interventions: Other: Potted Mint Plants

INTERVENTIONS:
Other: Potted Mint Plants — We will measure 2 indoor environments (living room and bedroom) for placing potted plants.

SUMMARY:
This study will recruit 60 subjects, in sum of 30 families. We will measure 2 indoor environments (living room and bedroom) for All-in-one monitoring the indoor air quality, in which collected culturable fungus and bacteria indoor to calculate colony forming unit (CFU). We will apply Kore Technology (MS-200) (Electron Ionization time-of-flight mass spectrometry, EI-TOF-MS) to measure the indoor volatile organic chemicals (VOCs) before intervention and perform repeated measurements of VOCs and the concentration of phytoncides before intervention and one week later after placing potted plants into indoor environments (living room and bedroom).

In conclusion, this study aims to investigate the clinical utility of potted mint plants in reducing indoor bacterial and fungal growth and indoor air pollution, and cardiovascular benefits. Furthermore, the possible application of indoor potted mint plant in antiviral influenza or pneumonia in the future.

DETAILED DESCRIPTION:
The contribution of air pollution is a very important public health issue for human health. Indoor air quality may have more influence on human health than outdoor air pollution. Previous studies indicate indoor air pollution which causes respiratory disease has been associated with cardiovascular disease. Besides, some studies showed that indoor CO2 concentration was positively correlated with virus detection and bacterial concentration in the air, and coagulase-negative staphylococci (CNS) was detected in many poorly ventilated indoor environments. Mint can release chemical substance to inhibit viruses and bacteria. Among the components, the menthol and terpineol induced vasodilation so as to reduce blood pressure. For the pilot study we have finished the qualitative and quantitative research in chemical components released by the mint.

Therefore, this study aims to evaluate the indoor air quality and the distribution of fungal and bacterial concentration in the indoor environment, analyze the effect of potted mint plants on indoor air quality, fungal and bacterial concentration, and explore the correlation between the intervention of potted mint plants and cardiovascular health.

This study will recruit 60 subjects, in sum of 30 families. We will measure 2 indoor environments (living room and bedroom) for All-in-one monitoring the indoor air quality, in which collected culturable fungus and bacteria indoor to calculate colony forming unit (CFU). We will apply Kore Technology (MS-200) (Electron Ionization time-of-flight mass spectrometry, EI-TOF-MS) to measure the indoor volatile organic chemicals (VOCs) before intervention and perform repeated measurements of VOCs and the concentration of phytoncides before intervention and one week later after placing potted plants into indoor environments (living room and bedroom).

Furthermore, we used matrix-assisted laser desorption ionization time of flight mass spectrometry (MALDI-TOF-MS) to identify microbiology; simultaneously, we record the outdoor environment and indoor ventilation. To assess subjects' cardiovascular health, we use DynaPulse to evaluate their cardiovascular function, and make them equipped with Holter electrocardiography (ECG) to continuously monitor the trend of heart rate variability (HRV) before and after intervention.

In conclusion, this study aims to investigate the clinical utility of potted mint plants in reducing indoor bacterial and fungal growth and indoor air pollution, and cardiovascular benefits. Furthermore, the possible application of indoor potted mint plant in antiviral influenza or pneumonia in the future.

ELIGIBILITY:
Inclusion Criteria:

* in the Department of Cardiology or inpatients at National Taiwan University Hospital
* aged 20-80
* live in the Greater Taipei area

Exclusion Criteria:

* The research subjects must agree to cooperate with the health assessment.
* serious brain, heart disease and mental illness
* uncomfortable reactions

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Improve Indoor Air Quality | one week

CONTACTS AND LOCATIONS:
Overall Officials: Su ta chen, PI, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Chung-Shan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided